CLINICAL TRIAL: NCT03060577
Title: An Open Label, Active Comparator Extension Trial to Assess the Effect of Long Term Dosing of Inclisiran and Evolocumab Given as Subcutaneous Injections in Participants With High Cardiovascular Risk and Elevated LDL-C (ORION-3)
Brief Title: An Extension Trial of Inclisiran in Participants With Cardiovascular Disease and High Cholesterol
Acronym: ORION-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-PCS-16-01; 2016-003815-37 (EudraCT Number)
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Atherosclerotic Cardiovascular Disease; Symptomatic Atherosclerosis; Type2 Diabetes; Familial Hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis; Hyperlipoproteinemia Type II | interventions — ALN-PCS; evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran-only (Experimental): Participants received subcutaneous injections of inclisiran 300 milligrams (mg) on Day 1 and every 180 days thereafter for up to 4 years.
  Interventions: Drug: Inclisiran
- Switching (Active Comparator): Participants received self-administered subcutaneous injections of evolocumab 140 mg on Day 1 and every 14 days thereafter until Day 336. Then, participants received subcutaneous injections of inclisiran 300 mg on Day 360 and every 180 days thereafter for up to 4 years.
  Interventions: Drug: Inclisiran; Drug: Evolocumab

INTERVENTIONS:
Drug: Inclisiran — Inclisiran is a synthetic, chemically modified small interfering ribonucleic acid (siRNA) targeting proprotein convertase subtilisin kexin type 9 (PCSK9) messenger ribonucleic acid (mRNA) with a covalently attached triantennary N-acetylgalactosamine (GalNAc) ligand.
  Other Names: ALN-PCSSC
Drug: Evolocumab — Evolocumab is a fully human monoclonal antibody that inhibits PCSK9.
  Other Names: REPATHA
  Arms: Switching

SUMMARY:
This clinical study was designed to assess the efficacy, safety, and tolerability of long-term dosing of inclisiran and evolocumab given as subcutaneous injections in participants with high cardiovascular risk and elevated low-density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
MDCO-PCS-16-01 (ORION-3) was a Phase II, open-label, multicenter, non-randomized, active comparator long term extension study. Total study duration was 4 years from first participant enrolled to the last subject completed. The study consisted of three study periods:

Screening Period: Participants completing study MDCO-PCS-15-01 (ORION-1) were screened for all inclusion and exclusion criteria of study ORION-3.

Treatment Period: Participants fulfilling all eligibility criteria of ORION-3 were enrolled. Participants who received inclisiran in ORION-1 received inclisiran sodium throughout this study up to 4 years (Group 1; Inclisiran-only arm), and participants who received placebo in ORION-1 received evolocumab as open-label comparator up to Day 336, and then transitioned to inclisiran on Day 360 and every 180 days thereafter for up to 4 years (Group 2; Switching arm).

Safety follow up: Participants were followed up for safety during 4 weeks after the last dose of study treatment. Including the Screening Period, the total study duration for a participant was up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of Study MDCO-PCS-15-01 and no contraindication to receiving inclisiran or evolocumab.
2. Willing and able to give written and informed consent before initiation of any study related procedures and willing to comply with all required study procedures.
3. Willing to self-inject.

Exclusion Criteria:

1. Any uncontrolled or serious disease, or any medical or surgical condition that may either interfere with participation in the clinical study and/or put the participant at significant risk (according to investigator's [or delegate's] judgment).
2. An underlying known disease or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate), might interfere with interpretation of the clinical study results.
3. Serious comorbid disease in which the life expectancy of the participant is shorter than the duration of the trial (for example, acute systemic infection, cancer, or other serious illnesses).
4. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver; unexplained alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation greater than 2 times upper limit of normal (ULN); or total bilirubin elevation greater than 1.5 times ULN at study entry visit.
5. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least two methods of contraception (for example, oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device) for the entire duration of the study. Exemptions from this criterion are

   * Women >2 years postmenopausal (defined as 1 year or longer since their last menstrual period) AND more than 55 years of age
   * Postmenopausal women (as defined above) and less than 55 years old with a negative pregnancy test within 24 hours of enrollment
   * Women who are surgically sterilized at least 3 months prior to enrollment
6. Males who are unwilling to use an acceptable method of birth control during the entire study period (that is, condom with spermicide).
7. Treatment with investigational medicinal products other than inclisiran or devices within 30 days or five half˗lives, whichever is longer.
8. Planned use of investigational medicinal products other than inclisiran or devices during the course of the study.
9. Participants with a history of a serious hypersensitivity reaction to evolocumab or any of the excipients
10. Previous or current treatment (within 90 days of study entry) with monoclonal antibodies directed towards PCSK9.
11. Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to:

    * Inappropriate for this study, including participants who are unable to communicate or to cooperate with the investigator.
    * Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study (including participants whose cooperation is doubtful due to drug abuse or alcohol dependency).
    * Unlikely to comply with the protocol requirements, instructions, and study-related restrictions (for example, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study).
    * Involved with, or a relative of, someone directly involved in the conduct of the study.
    * Any known cognitive impairment (for example, Alzheimer's Disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kausik Ray, MD, Principal Investigator — Imperial College London
Locations (49):
- United States (7):
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Greenville, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Richmond, Virginia
- Canada (10):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Québec
  - Novartis Investigative Site, St. Johns
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Munich
- Netherlands (13):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Rotterdam, The Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Goes
  - Novartis Investigative Site, Hoogeveen
  - Novartis Investigative Site, Hoogezand
  - Novartis Investigative Site, Hoorn
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Venlo
  - Novartis Investigative Site, Zwijndrecht
- United Kingdom (14):
  - Novartis Investigative Site, Fowey, Cornwall
  - Novartis Investigative Site, Liskeard, Cornwall
  - Novartis Investigative Site, Penzance, Cornwall
  - Novartis Investigative Site, St Austell, Cornwall
  - Novartis Investigative Site, Torpoint, Cornwall
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, High Wycombe
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle Upon Tyme
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Worcester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ray KK, Troquay RPT, Visseren FLJ, Leiter LA, Scott Wright R, Vikarunnessa S, Talloczy Z, Zang X, Maheux P, Lesogor A, Landmesser U. Long-term efficacy and safety of inclisiran in patients with high cardiovascular risk and elevated LDL cholesterol (ORION-3): results from the 4-year open-label extension of the ORION-1 trial. Lancet Diabetes Endocrinol. 2023 Feb;11(2):109-119. doi: 10.1016/S2213-8587(22)00353-9. Epub 2023 Jan 5. PMID 36620965
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 51 sites in 5 countries.
Pre-assignment Details: After completion of study MDCO-PCS-15-01, participants were screened to fulfill all inclusion and exclusion criteria.
Groups:
- Inclisiran-only: Participants received subcutaneous injections of inclisiran 300 milligrams (mg) on Day 1 and every 180 days thereafter up to Year 4.
- Switching: Participants received self-administered subcutaneous injections of evolocumab 140 mg on Day 1 and every 14 days thereafter until Day 336. Then, participants received subcutaneous injections of inclisiran 300 mg on Day 360 and every 180 days thereafter up to Year 4.
Period: Overall Study
Arm/Group | Inclisiran-only | Switching
Started (All enrolled participants) | 290 | 92
Safety Analysis Set (All enrolled participants who received at least one dose of study treatment) | 284 | 90
Completed | 233 | 80
Not Completed | 57 | 12
Not completed — Withdrawal by Subject | 25 | 5
Not completed — Physician Decision | 4 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 7 | 1
Not completed — Adverse Event | 9 | 1
Not completed — Inclusion/Exclusion | 1 | 0
Not completed — Other | 8 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran-only | Switching | Total
Number analyzed (Participants) | 290 | 92 | 382
Age, Continuous [Mean (Standard Deviation); unit: Year] | 63.3 (11.14) | 61.9 (10.56) | 63.0 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 37 | 139
  Male | 188 | 55 | 243
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 7 | 22
  Not Hispanic or Latino | 275 | 85 | 360
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline of the ORION-1 Study to Day 210 in ORION-3 (Inclisiran Arm)
Description: Percent Change in LDL-C (beta-quantification) from baseline of the ORION-1 Study to Day 210 in ORION-3. A negative percentage score represents a reduction in LDL-C. Change is relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Day 210 (ORION-3) (up to 570 days total)
Population: The overall number of participants analyzed includes all participants in the Safety Analysis Set of the Inclisiran-only arm with evaluable data for the endpoint.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
Percentage Change | -47.48 [-50.69 to -44.27]

2. Secondary Outcome: Percentage Change in LDL-C From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Percent Change in LDL-C (beta-quantification) from baseline of the ORION-1 Study overtime in ORION-3. A negative percentage score represents a reduction in LDL-C. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 360, 720, 1080 and 1440 (ORION-3) (up to 390, 720, 1080, 1440 and 1800 days total, respectively)
Population: The overall number of participants and the number analyzed per row represents participants in the Safety Analysis set of the Inclisiran-only arm with evaluable data at each time point.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
Percentage Change
  Day 30 | -49.43 [-52.27 to -46.58]
  Day 360: number analyzed (Participants) | 269
  Day 360 | -37.14 [-40.95 to -33.32]
  Day 720: number analyzed (Participants) | 253
  Day 720 | -38.43 [-41.75 to -35.11]
  Day 1080: number analyzed (Participants) | 225
  Day 1080 | -51.07 [-54.75 to -47.39]
  Day 1440: number analyzed (Participants) | 232
  Day 1440 | -46.74 [-50.71 to -42.78]

3. Secondary Outcome: Absolute Change in LDL-C From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Absolute Change in LDL-C (beta-quantification) from baseline of the ORION-1 Study overtime in ORION-3. A negative score represents a reduction in LDL-C. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
mg/dL
  Day 30 | -62.51 [-66.76 to -58.25]
  Day 360: number analyzed (Participants) | 269
  Day 360 | -47.96 [-52.56 to -43.35]
  Day 720: number analyzed (Participants) | 253
  Day 720 | -49.44 [-54.25 to -44.64]
  Day 1080: number analyzed (Participants) | 225
  Day 1080 | -63.34 [-68.76 to -57.92]
  Day 1440: number analyzed (Participants) | 232
  Day 1440 | -60.04 [-65.81 to -54.27]

4. Secondary Outcome: Percentage Change in PCSK9 Levels From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Percent Change in PCSK9 from baseline of the ORION-1 Study overtime in ORION-3. A negative percentage score represents a reduction in PCSK9. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 360, 720 and 1440 (ORION-3) (up to 390, 720, 1080 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
Percentage Change
  Day 30 | -71.80 [-73.17 to -70.44]
  Day 360: number analyzed (Participants) | 271
  Day 360 | -63.79 [-65.79 to -61.80]
  Day 720: number analyzed (Participants) | 253
  Day 720 | -62.17 [-64.46 to -59.88]
  Day 1440: number analyzed (Participants) | 228
  Day 1440 | -69.54 [-71.19 to -67.89]

5. Secondary Outcome: Absolute Change in PCSK9 Levels From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Absolute Change in PCSK9 from baseline of the ORION-1 Study overtime in ORION-3. A negative score represents a reduction in PCSK9. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 360, 720 and 1440 (ORION-3) (up to 390, 720, 1080 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ug/L
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
ug/L
  Day 30 | -314.07 [-328.69 to -299.45]
  Day 360: number analyzed (Participants) | 271
  Day 360 | -280.88 [-295.71 to -266.06]
  Day 720: number analyzed (Participants) | 253
  Day 720 | -275.78 [-291.91 to -259.64]
  Day 1440: number analyzed (Participants) | 228
  Day 1440 | -314.34 [-331.22 to -297.46]

6. Secondary Outcome: Percentage Change in Triglycerides From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Percent Change in Triglycerides from baseline of the ORION-1 Study overtime in ORION-3. A negative percentage score represents a reduction in Triglycerides. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 210 and 1440 (ORION-3) (up to 390, 570 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
Percentage Change
  Day 30 | -1.71 [-6.42 to 3.00]
  Day 210 | -3.35 [-9.12 to 2.41]
  Day 1440: number analyzed (Participants) | 232
  Day 1440 | 0.73 [-8.23 to 9.69]

7. Secondary Outcome: Absolute Change in Triglycerides From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Absolute Change in Triglycerides from baseline of the ORION-1 Study overtime in ORION-3. A negative score represents a reduction in Triglycerides. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 210 and 1440 (ORION-3) (up to 390, 570 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
mg/dL
  Day 30 | -14.61 [-22.15 to -7.08]
  Day 210 | -11.96 [-23.78 to -0.14]
  Day 1440: number analyzed (Participants) | 232
  Day 1440 | -14.83 [-25.75 to -3.90]

8. Secondary Outcome: Percentage Change in Apolipoprotein B From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Percent Change in Apolipoprotein B from baseline of the ORION-1 Study overtime in ORION-3. A negative percentage score represents a reduction in Apolipoprotein B. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 210 and 1440 (ORION-3) (up to 390, 570 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
Percentage Change
  Day 30 | -40.43 [-42.57 to -38.29]
  Day 210 | -36.65 [-39.06 to -34.23]
  Day 1440: number analyzed (Participants) | 226
  Day 1440 | -33.66 [-37.18 to -30.15]

9. Secondary Outcome: Absolute Change in Apolipoprotein B From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Absolute Change in Apolipoprotein B from baseline of the ORION-1 Study overtime in ORION-3. A negative score represents a reduction in Apolipoprotein B. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 210 and 1440 (ORION-3) (up to 390, 570 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
mg/dL
  Day 30 | -42.63 [-45.22 to -40.04]
  Day 210 | -38.36 [-41.19 to -35.54]
  Day 1440: number analyzed (Participants) | 226
  Day 1440 | -36.26 [-40.01 to -32.52]

10. Secondary Outcome: Percentage Change in Lipoprotein-a From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Percent Change in Lipoprotein-a from baseline of the ORION-1 Study overtime in ORION-3. A negative percentage score represents a reduction in Lipoprotein-a. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 210 and 1440 (ORION-3) (up to 390, 570 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
Percentage Change
  Day 30 | -15.88 [-19.48 to -12.28]
  Day 210 | 9.29 [4.42 to 14.16]
  Day 1440: number analyzed (Participants) | 225
  Day 1440 | -5.24 [-9.86 to -0.61]

11. Secondary Outcome: Absolute Change in Lipoprotein-a From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Absolute Change in Lipoprotein-a from baseline of the ORION-1 Study overtime in ORION-3. A negative score represents a reduction in Lipoprotein-a. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 210 and 1440 (ORION-3) (up to 390, 570 and 1800 days total, respectively)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 277
nmol/L
  Day 30 | -8.52 [-12.25 to -4.79]
  Day 210 | -4.94 [-8.67 to -1.20]
  Day 1440: number analyzed (Participants) | 225
  Day 1440 | -4.78 [-9.63 to 0.06]

12. Secondary Outcome: Number of Participants With ≥50% LDL-C Reduction From Baseline of the ORION-1 Study (Inclisiran Arm)
Description: Number of Participants with ≥50% LDL-C (beta-quantification) Reduction from baseline of the ORION-1 Study overtime in ORION-3. Changes are relative to ORION-1 Baseline, which is defined as the last available record prior to first study drug administration in ORION-1.
Time Frame: Baseline (ORION-1) and Days 30, 360, 720 and 1440 (ORION-3) (up to 390, 720, 1080 and 1800 days total, respectively)
Population: The overall number of participants and the number analyzed includes all participants in the Safety Analysis set of the Inclisiran-only arm. The number analyzed per row represents participants with evaluable data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 284
Participants
  Day 30 | 161
  Day 360: number analyzed (Participants) | 271
  Day 360 | 99
  Day 720: number analyzed (Participants) | 255
  Day 720 | 97
  Day 1440: number analyzed (Participants) | 234
  Day 1440 | 122

13. Secondary Outcome: Number of Participants Reaching on Treatment LDL-C Levels of <25 mg/dL, <50 mg/dL, <70 mg/dL, and <100 mg/dL (Inclisiran Arm)
Description: Individual responsiveness to inclisiran is defined as the number of Participants Reaching on Treatment LDL-C Levels of <25 mg/dL, <50 mg/dL, <70 mg/dL, and <100 mg/dL at any time point.
Time Frame: From the start of treatment in ORION-3 to 90 days after end of treatment, assessed up to maximum duration of 4 years
Population: The overall number of participants and the number analyzed includes all participants in the Safety Analysis set of the Inclisiran-only arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran-only
Number analyzed (Participants) | 284
Participants
  LDL-C level <25 mg/dL | 82
  LDL-C level <50 mg/dL | 175
  LDL-C level <70 mg/dL | 225
  LDL-C level <100 mg/dL | 265

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment in ORION-3 up to end of study visit, assessed up to maximum duration of 4 years.
Groups:
- Inclisiran Only Arm: Participants received subcutaneous injections of inclisiran 300 milligrams (mg) on Day 1 and every 180 days thereafter up to Year 4.
- Switching Arm up to Day 360 Visit: Participants received self-administered subcutaneous injections of evolocumab 140 mg on Day 1 and every 14 days thereafter until Day 336.
- Switching Arm After Day 360 Visit: Participants received subcutaneous injections of inclisiran 300 mg on Day 360 and every 180 days thereafter up to Year 4.
Arm/Group | Inclisiran Only Arm | Switching Arm up to Day 360 Visit | Switching Arm After Day 360 Visit
All-Cause Mortality (participants affected / at risk) | 7/284 | 0/90 | 1/87
Serious Adverse Events (participants affected / at risk) | 104/284 | 16/90 | 30/87
Other Adverse Events (participants affected / at risk) | 271/284 | 78/90 | 77/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran Only Arm (N=284) | Switching Arm up to Day 360 Visit (N=90) | Switching Arm After Day 360 Visit (N=87)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 1 | 2
Angina pectoris (Cardiac disorders) | 7 | 0 | 1
Angina unstable (Cardiac disorders) | 5 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 4 | 1 | 3
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 1 | 1
Vascular stent restenosis (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 6 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Infected bite (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Pulse abnormal (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hodgkin's disease stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Testicular seminoma (pure) stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 0 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urethral perforation (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Giant cell arteritis (Vascular disorders) | 0 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 2
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran Only Arm (N=284) | Switching Arm up to Day 360 Visit (N=90) | Switching Arm After Day 360 Visit (N=87)
Anaemia (Blood and lymphatic system disorders) | 6 | 4 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
White blood cell disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 17 | 4 | 5
Aortic valve incompetence (Cardiac disorders) | 3 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 10 | 0 | 2
Atrial flutter (Cardiac disorders) | 2 | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 3 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Bundle branch block left (Cardiac disorders) | 3 | 0 | 0
Bundle branch block right (Cardiac disorders) | 3 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 1
Coronary artery aneurysm (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 4 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Dilatation atrial (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 7 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Right ventricular dilatation (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 2 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 2 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 4 | 1 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 2 | 1 | 3
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 9 | 1 | 3
Vertigo positional (Ear and labyrinth disorders) | 2 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 4 | 1 | 2
Thyroid cyst (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 15 | 0 | 3
Chalazion (Eye disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Corneal erosion (Eye disorders) | 1 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 2 | 0 | 0
Dry eye (Eye disorders) | 4 | 0 | 3
Entropion (Eye disorders) | 0 | 1 | 0
Epiretinal membrane (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 1
Glaucoma (Eye disorders) | 1 | 1 | 0
Iritis (Eye disorders) | 1 | 0 | 0
Lacrimal mucocoele (Eye disorders) | 1 | 0 | 0
Lacrimation decreased (Eye disorders) | 1 | 0 | 0
Macular degeneration (Eye disorders) | 4 | 1 | 1
Macular hole (Eye disorders) | 0 | 0 | 1
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 1
Meibomianitis (Eye disorders) | 1 | 0 | 0
Metamorphopsia (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1
Retinal artery embolism (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 1
Retinopathy hypertensive (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 1 | 2
Visual impairment (Eye disorders) | 1 | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 10 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 4 | 3
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 2 | 0 | 0
Buccal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 15 | 5 | 5
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 3 | 9
Diverticulum (Gastrointestinal disorders) | 5 | 1 | 4
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal scarring (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2 | 5
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 2 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 6 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 2 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 9 | 1 | 3
Levator syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Malpositioned teeth (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 18 | 3 | 6
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic steatosis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Salivary gland disorder (Gastrointestinal disorders) | 1 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 8 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 2 | 1
Adverse drug reaction (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 5 | 0 | 0
Chest discomfort (General disorders) | 5 | 0 | 1
Chest pain (General disorders) | 6 | 1 | 1
Chills (General disorders) | 2 | 0 | 1
Complication of device insertion (General disorders) | 0 | 1 | 0
Crepitations (General disorders) | 1 | 0 | 0
Cyst (General disorders) | 2 | 0 | 1
Discomfort (General disorders) | 0 | 1 | 0
Drug intolerance (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 23 | 3 | 10
Feeling abnormal (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 15 | 2 | 3
Injection site bruising (General disorders) | 4 | 4 | 3
Injection site discolouration (General disorders) | 3 | 0 | 0
Injection site erythema (General disorders) | 12 | 0 | 3
Injection site haematoma (General disorders) | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 2 | 1 | 0
Injection site oedema (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 12 | 0 | 4
Injection site paraesthesia (General disorders) | 0 | 0 | 1
Injection site pruritus (General disorders) | 1 | 0 | 0
Injection site rash (General disorders) | 8 | 0 | 1
Injection site reaction (General disorders) | 16 | 2 | 4
Injection site urticaria (General disorders) | 1 | 0 | 0
Injection site vesicles (General disorders) | 0 | 0 | 1
Injection site warmth (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 1
Medical device complication (General disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 13 | 1 | 4
Oedema peripheral (General disorders) | 11 | 2 | 6
Pain (General disorders) | 2 | 0 | 0
Peripheral swelling (General disorders) | 4 | 1 | 1
Polyp (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0
Vessel puncture site induration (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 7 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 5 | 0 | 2
Allergy to animal (Immune system disorders) | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 2 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0
Food allergy (Immune system disorders) | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Mite allergy (Immune system disorders) | 1 | 0 | 0
Rubber sensitivity (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 2 | 2
Abscess (Infections and infestations) | 1 | 0 | 0
Abscess of eyelid (Infections and infestations) | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Balanitis candida (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 15 | 3 | 4
COVID-19 (Infections and infestations) | 3 | 0 | 2
Candida infection (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 3 | 0 | 1
Corneal infection (Infections and infestations) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 3 | 0 | 0
Cystitis (Infections and infestations) | 5 | 2 | 6
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 5 | 2 | 2
Ear infection (Infections and infestations) | 1 | 1 | 5
Ear lobe infection (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
External ear cellulitis (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 3 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 5 | 0 | 0
Fungal skin infection (Infections and infestations) | 3 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 12 | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 8 | 2 | 2
Genital herpes simplex (Infections and infestations) | 1 | 0 | 0
Genital infection fungal (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 3
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 12 | 1 | 3
Hordeolum (Infections and infestations) | 5 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 36 | 6 | 10
Kidney infection (Infections and infestations) | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 11 | 1 | 1
Mastitis (Infections and infestations) | 1 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 55 | 6 | 13
Onychomycosis (Infections and infestations) | 4 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 2 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 1
Oral infection (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 3 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Perichondritis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 0 | 3
Pneumonia (Infections and infestations) | 2 | 2 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1
Retinitis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 0
Root canal infection (Infections and infestations) | 1 | 0 | 0
Sebaceous gland infection (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 10 | 3 | 3
Skin infection (Infections and infestations) | 3 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 2 | 0 | 1
Tooth infection (Infections and infestations) | 3 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 24 | 1 | 5
Urethritis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 37 | 6 | 7
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 2 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 2 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 0
Wound infection (Infections and infestations) | 2 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 5 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 15 | 2 | 3
Epicondylitis (Injury, poisoning and procedural complications) | 2 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 24 | 1 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 3 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 4 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 0 | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 3 | 1
Lip injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 4 | 0 | 0
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1 | 1
Product dispensing error (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Reactive gastropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 6 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 3
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 5 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 6 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 3 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Wrong dose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 10 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood folate decreased (Investigations) | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 5 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 2 | 0 | 0
Blood pressure increased (Investigations) | 1 | 1 | 1
Blood sodium decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 2 | 0 | 0
Blood uric acid decreased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 5 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Carbohydrate antigen 19-9 increased (Investigations) | 1 | 0 | 0
Carcinoembryonic antigen increased (Investigations) | 2 | 0 | 0
Cardiac murmur (Investigations) | 1 | 1 | 0
Carotid bruit (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 2 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 2 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 1
Heart rate decreased (Investigations) | 1 | 0 | 0
Heart rate irregular (Investigations) | 3 | 0 | 0
Hepatic enzyme increased (Investigations) | 9 | 0 | 2
International normalised ratio increased (Investigations) | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1
Lipoprotein (a) increased (Investigations) | 1 | 0 | 0
Lipoprotein increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 3 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Mean cell volume increased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 2 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 1
Pulse absent (Investigations) | 1 | 0 | 0
QRS axis abnormal (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 0 | 0
Sinus rhythm (Investigations) | 1 | 0 | 0
Spirometry abnormal (Investigations) | 1 | 0 | 0
Streptococcus test positive (Investigations) | 1 | 0 | 0
Thyroid function test abnormal (Investigations) | 1 | 0 | 0
Troponin T increased (Investigations) | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 2 | 0 | 0
Vitamin B12 decreased (Investigations) | 1 | 0 | 0
Vitamin D decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 2
Weight increased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 32 | 0 | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 | 0 | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 2 | 0
Gout (Metabolism and nutrition disorders) | 12 | 1 | 5
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 2 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 7 | 0 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 10 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 1 | 3
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 1 | 13
Bone atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 6 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 2 | 6
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 1 | 6
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Shoulder deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 0 | 3
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 2 | 0 | 0
Burning sensation (Nervous system disorders) | 2 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 2 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 3 | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Cluster headache (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 3 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 24 | 4 | 5
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 21 | 8 | 7
Hypoaesthesia (Nervous system disorders) | 4 | 2 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 3 | 0 | 0
Migraine (Nervous system disorders) | 2 | 1 | 2
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Muscle tension dysphonia (Nervous system disorders) | 1 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 2
Occipital neuralgia (Nervous system disorders) | 0 | 1 | 1
Ophthalmic migraine (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 7 | 1 | 3
Parkinson's disease (Nervous system disorders) | 2 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Piriformis syndrome (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 5 | 1 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 2
Sciatica (Nervous system disorders) | 3 | 1 | 3
Sensory loss (Nervous system disorders) | 3 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 1
Syncope (Nervous system disorders) | 4 | 0 | 2
Taste disorder (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 3 | 0 | 0
Vascular dementia (Nervous system disorders) | 2 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
Prosthetic cardiac valve failure (Product Issues) | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Burnout syndrome (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 12 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 1 | 0
Emotional distress (Psychiatric disorders) | 1 | 0 | 0
Fear (Psychiatric disorders) | 1 | 0 | 0
Indifference (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 10 | 1 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 1
Seasonal affective disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Albuminuria (Renal and urinary disorders) | 1 | 0 | 0
Bladder cyst (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 3 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 9 | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 2 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 2 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 3 | 0 | 0
Myoglobinuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 4 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 4 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 3 | 1 | 1
Ureteral disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 0
Urinary tract discomfort (Renal and urinary disorders) | 1 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 0 | 3
Breast disorder female (Reproductive system and breast disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 3 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0 | 0
Penile erythema (Reproductive system and breast disorders) | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 1
Spermatocele (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 1 | 5
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 5
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Actinic elastosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2 | 2
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 2 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 2 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 6 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Xanthoma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0 | 2
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 2 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 42 | 2 | 17
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 6 | 0 | 1
Intermittent claudication (Vascular disorders) | 3 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 2 | 0 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Varicophlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03060577/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03060577/SAP_001.pdf